CLINICAL TRIAL: NCT06833073
Title: A Phase 2 Open-label Randomized Study of V940 in Combination With BCG Versus BCG Monotherapy in Participants With High-risk Non-muscle Invasive Bladder Cancer (INTerpath-011)
Brief Title: A Clinical Study of Intismeran Autogene (V940) and BCG in People With Bladder Cancer (V940-011/INTerpath-011)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V940-011; 2024-517335-46-00 (Registry Identifier: EU CT); U1111-1312-0572 (Registry Identifier: UTN); INTerpath-011 (Other: MSD); V940-011 (Other: MSD)
Record Dates: First submitted 2025-02-04; First posted 2025-02-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Carcinoma in Situ
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Carcinoma in Situ | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: Participants allocated to receive BCG will be randomized 1:1 to the intismeran autogene+BCG arm and the BCG arm (Cohort A).
  Participants allocated to receive intismeran autogene monotherapy will be allocated to the single intismeran autogene monotherapy arm (Cohort B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intismeran autogene + BCG (Experimental): Participants in Cohort A receive 1 mg of intismeran autogene via intramuscular (IM) injection every 3 weeks (Q3W) for 9 doses. Participants also receive 50 mg of TICE® BCG once weekly for 6 weeks, then once weekly on weeks 13-15, 25-27, 49-51, and 73-75.
  Interventions: Biological: Intismeran autogene; Biological: BCG
- BCG (Active Comparator): Participants in Cohort A receive 50 mg of TICE® BCG once weekly for 6 weeks, then once weekly on weeks 13-15, 25-27, 49-51, and 73-75.
  Interventions: Biological: BCG
- Intismeran autogene (Experimental): Participants in Cohort B receive 1 mg of intismeran autogene via intramuscular (IM) injection every 3 weeks (Q3W) for 9 doses.
  Interventions: Biological: Intismeran autogene

INTERVENTIONS:
Biological: Intismeran autogene — IM injection
  Other Names: mRNA-4157; V940
  Arms: Intismeran autogene; Intismeran autogene + BCG
Biological: BCG — Intravesicular instillation. BCG is a preparation of Bacillus Calmette-Guerin.
  Other Names: BCG Live; TICE®; TheraCys®
  Arms: BCG; Intismeran autogene + BCG

SUMMARY:
Researchers are looking for new ways to treat people with high-risk non-muscle invasive bladder cancer (HR NMIBC). NMIBC is cancer in the tissue that lines the inside of the bladder but has not spread to the bladder muscle or outside of the bladder. High-risk means NMIBC may have a high chance of getting worse or coming back after treatment. HR NMIBC can also include carcinoma in situ (CIS). CIS is bladder cancer that appears flat and is only in the inner layer (surface) of the bladder. CIS is not raised and is not growing toward the center of the bladder.

The standard treatment for HR NMIBC is a procedure to remove the tumor called transurethral resection of the bladder tumor (TURBT) followed by Bacillus Calmette-Guerin (BCG). Standard treatment is something that is considered the first line of treatment for a condition. BCG is an immunotherapy, which is a treatment that helps the immune system fight cancer. However, BCG may not work to treat HR NMIBC in some people. Researchers want to learn if adding intismeran autogene, the study treatment, to standard treatment can help treat HR NMIBC. Intismeran autogene is designed to help a person's immune system attack their specific cancer.

The goal of this study are to learn if people who receive V940 with BCG live longer and without the cancer growing, spreading, or coming back compared to people who receive BCG alone.

DETAILED DESCRIPTION:
As of Amendment 03 (effective 01/05/2026), outcome measures associated with the Intismeran autogene Monotherapy Arm (Cohort B) are no longer considered primary or secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Is an individual whose most recent TURBT was performed within 12 weeks before randomization/allocation and showed BICR-confirmed high-risk NMIBC histology

Cohort A:

* Has high-risk non-muscle invasive (HG Ta, T1, and/or CIS) UC of the bladder
* Is BCG-naïve defined as either having never received BCG or having received BCG more than 2 years before high-risk NMIBC recurrence. Recurrence must be at least 24 months from the last exposure to BCG with evidence of complete response during the 2-year period post BCG

Cohort B:

* Has CIS +/-papillary non-muscle invasive UC of the bladder
* Is ineligible for, or refusing, any IVESIC therapy
* Is either BCG-naïve (as defined above) or BCG-exposed but did not receive protocol-specified minimum dosing of BCG and experienced recurrence of high-risk NMIBC within 2 years of the last dose of BCG
* Human immunodeficiency virus (HIV)-infected individuals must have well controlled HIV on antiretroviral therapy (ART)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of or concurrent locally-advanced (ie, T2, T3, T4) or metastatic UC
* Has concurrent extravesical (ie, urethra, ureter, renal pelvis) non-muscle invasive UC or a history of extravesical non-muscle invasive UC that recurred within the last 2 years, with certain exceptions
* Has a known additional malignancy that is progressing or has required active treatment within the last 3 years
* Has had a myocardial infarction within 6 months of randomization/allocation
* Has received any systemic anticancer therapy including investigational agents within 4 weeks before randomization/allocation
* Has received prior treatment with a cancer vaccine
* Has immunodeficiency or is receiving chronic systemic steroid therapy
* Has active autoimmune disease that has required systemic treatment in the last 2 years
* Has any contraindication to IV contrast and gadolinium or is otherwise unable to have imaging with either computerized tomography urogram (CTU) or Magnetic resonance urography (MRU)

Cohort A:

* Has current active tuberculosis
* Has a known history of HIV infection

Cohort B:

- HIV-infected individuals with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2031-09-03 (Estimated); Study Completion 2031-09-03 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Event-free Survival (EFS) | Up to approximately 5 years
  EFS is defined as the time from randomization to any of the following events, as determined by blinded independent central review (BICR) where applicable: High-grade (HG) non-invasive papillary carcinoma (Ta) or carcinoma in situ (CIS) in the bladder at the 24-week assessment or later; Any T1 stage disease in the bladder; Any T2 stage or greater in the bladder, including transurethral prostate stromal invasion of urothelial carcinoma (UC); High-risk disease (defined as HG Ta, CIS, ≥T1) of the urethra or upper tract (ureters, renal pelvis); Metastatic UC [defined as regional lymph node metastasis of UC (stage N1 or greater), or distant lymph node or visceral metastasis of UC (stage M1)]; Or death due to any cause. The EFS for BCG-treated participants will be presented.

SECONDARY OUTCOMES:
Cohort A: 12-Month Event-free Survival (EFS) | Up to approximately 12 months
  EFS is defined as the time from randomization to any of the following events, as determined by BICR where applicable: HG Ta or CIS in the bladder at the 24-week assessment or later; Any T1 stage disease in the bladder; Any T2 stage or greater in the bladder, including transurethral prostate stromal invasion of UC; High-risk disease (defined as HG Ta, CIS, ≥T1) of the urethra or upper tract (ureters, renal pelvis); Metastatic UC [defined as regional lymph node metastasis of UC (stage N1 or greater), or distant lymph node or visceral metastasis of UC (stage M1)]; Or death due to any cause. The EFS at 12 months for BCG-treated participants will be presented.
Cohort A: 24-Month Event-free Survival (EFS) | Up to approximately 24 months
  EFS is defined as the time from randomization to any of the following events, as determined by BICR where applicable: HG Ta or CIS in the bladder at the 24-week assessment or later; Any T1 stage disease in the bladder; Any T2 stage or greater in the bladder, including transurethral prostate stromal invasion of UC; High-risk disease (defined as HG Ta, CIS, ≥T1) of the urethra or upper tract (ureters, renal pelvis); Metastatic UC [defined as regional lymph node metastasis of UC (stage N1 or greater), or distant lymph node or visceral metastasis of UC (stage M1)]; Or death due to any cause. The EFS at 24 months for BCG-treated participants will be presented.
Cohort A: Recurrence-free Survival (RFS) | Up to approximately 5 years
  RFS is defined as the time from randomization to any of the following events, as determined by BICR where applicable: HG Ta or CIS in the bladder at the 24-week assessment or later; Any T1 stage disease in the bladder; Any T2 stage or greater in the bladder, including transurethral prostate stromal invasion of UC; High-risk disease (defined as HG Ta, CIS, ≥T1) of the urethra or upper tract (ureters, renal pelvis); Metastatic UC [defined as regional lymph node metastasis of UC (stage N1 or greater), or distant lymph node or visceral metastasis of UC (stage M1)]; Death due to any cause; or any other UC recurrence including low-grade (LG) Ta at any timepoint as well as HG Ta or CIS in the bladder before the 24-week assessment. The RFS will be presented.
Cohort A: Disease-specific Survival (DSS) | Up to approximately 5 years
  DSS is defined as the time from randomization to death due to bladder cancer. The DSS will be presented.
Cohort A: Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause.
Cohort A: 12 Month Overall Survival Rate (OSR) | Up to approximately 12 months
  OSR is defined as the percentage of participants who are alive at 12 months. The 12 month OSR for BCG-treated participants will be presented.
Cohort A: 24 Month Overall Survival Rate (OSR) | Up to approximately 24 months
  OSR is defined as the percentage of participants who are alive at 24 months. The 24 month OSR for BCG-treated participants will be presented.
Cohort A: Complete Response Rate (CRR) | Up to approximately 5 years
  CRR is defined as the percentage of participants who achieve a Complete Response (CR) defined as the absence of all of the following as determined by BICR using urine cytology, biopsy, and radiology assessments as applicable, and local cystoscopy evaluation: High-risk non-muscle invasive UC (defined as HG Ta, CIS, or any T1 disease of the bladder, urethra, or upper tract [ureters, renal pelvis]); Any T2 or greater in the bladder, including transurethral prostate stromal invasion of UC; Metastatic UC [defined as regional lymph node metastasis of UC (N1 or greater), or distant lymph node or visceral metastasis of UC (M1)]. The CRR for BCG-treated participants will be presented.
Cohort A: Duration of Response (DOR) | Up to approximately 5 years
  For participants who achieve a Complete Response (CR: the absence of all of the following as determined by BICR using urine cytology, biopsy, and radiology assessments as applicable, and local cystoscopy evaluation: High-risk non-muscle invasive UC (defined as HG Ta, CIS, or any T1 disease of the bladder, urethra, or upper tract [ureters, renal pelvis]); Any T2 or greater in the bladder, including transurethral prostate stromal invasion of UC; Metastatic UC [defined as regional lymph node metastasis of UC (N1 or greater), or distant lymph node or visceral metastasis of UC (M1)]), DOR is defined as the time from first documented CR to the first occurrence of any of the following: High-risk non-muscle invasive UC; muscle-invasive bladder cancer (MIBC) or locally-advanced or metastatic UC; Or death due to any cause. DOR as assessed by BICR will be presented.
Cohort A: Time to Cystectomy | Up to approximately 5 years
  Time to cystectomy, defined as the time from randomization to the date of cystectomy, will be presented for BCG-treated participants.
Cohort A: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 21 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE in the study will be presented.
Cohort A: Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 18 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue the study intervention due to an AE in the study will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (87):
- United States (20):
  - Michael G Oefelein Clinical Trials ( Site 0138), Bakersfield, California
  - Genesis Research, LLC ( Site 0141), Los Alamitos, California
  - USC Norris Comprehensive Cancer Center ( Site 0123), Los Angeles, California
  - Genesis Healthcare-Torrance ( Site 0140), Torrance, California
  - Genesis Research LLC ( Site 0118), Torrance, California
  - Urology Associates ( Site 0144), Littleton, Colorado
  - Urological Research Network ( Site 0133), Hialeah, Florida
  - Associated Urological Specialists - Chicago Ridge ( Site 0139), Chicago Ridge, Illinois
  - Southern Urology, LLC ( Site 0145), Lafayette, Louisiana
  - University of Missouri Health Care ( Site 0126), Columbia, Missouri
  - NHO Revive Research Institute, LLC ( Site 0137), Lincoln, Nebraska
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0111), New York, New York
  - TriState Urologic Services PSC Inc. dba The Urology Group ( Site 0122), Cincinnati, Ohio
  - OHSU Knight Cancer Institute - South Waterfront ( Site 0110), Portland, Oregon
  - MidLantic Urology ( Site 0102), Bala-Cynwyd, Pennsylvania
  - The Conrad Pearson Clinic ( Site 0143), Germantown, Tennessee
  - Texas Oncology-Austin Central ( Site 0107), Austin, Texas
  - Urology Austin, PLLC ( Site 0109), Austin, Texas
  - Urology of Virginia ( Site 0125), Virginia Beach, Virginia
  - University of Washington - Fred Hutchinson Cancer Center ( Site 0100), Seattle, Washington
- Argentina (7):
  - Hospital Italiano de Buenos Aires ( Site 0307), CABA, Buenos Aires
  - Instituto Alexander Fleming ( Site 0306), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar dle Plata ( Site 0305), Mar del Plata, Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés ( Site 0303), Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos ( Site 0304), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 0300), Rosario, Santa Fe Province
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0301), La Rioja
- Australia (2):
  - Macquarie University ( Site 1801), Macquarie University, New South Wales
  - Fiona Stanley Hospital ( Site 1803), Perth, Western Australia
- Brazil (4):
  - Instituto do Câncer e Transplante de Curitiba ( Site 0402), Curitiba, Paraná
  - Hospital de Clínicas de Passo Fundo ( Site 0406), Passo Fundo, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 0400), Barretos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0410), São Jose Do Rio Preto, São Paulo
- Canada (2):
  - The Moncton Hospital-Oncology ( Site 0200), Moncton, New Brunswick
  - CIUSSS de l'Estrie-CHUS ( Site 0204), Sherbrooke, Quebec
- Chile (6):
  - Oncocentro Valdivia ( Site 0507), Valdivia, Los Ríos Region
  - FALP ( Site 0500), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0502), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0501), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS ( Site 0505), Viña del Mar, Región de Valparaíso
  - Bradford Hill Norte ( Site 0503), Antofagasta
- Colombia (5):
  - Instituto de Cancerología ( Site 0600), Medellín, Antioquia
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 0603), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 0601), Montería, Departamento de Córdoba
  - Oncólogos del Occidente S.A.S. - Sede Pereira ( Site 0604), Pereira, Risaralda Department
  - Clínica Imbanaco S.A.S ( Site 0602), Cali, Valle del Cauca Department
- Herlev and Gentofte Hospital ( Site 3101), Herlev, Capital Region, Denmark
- France (5):
  - CHU Dijon Bourgogne ( Site 0802), Dijon, Cote-d Or
  - Bordeaux University Hospital - Pellegrin ( Site 0806), Bordeaux, Gironde
  - CHU de Rouen- urology ( Site 0803), Rouen, Haute-Normandie
  - Hôpital Foch-Urology department ( Site 0801), Suresnes, Hauts-de-Seine
  - Hôpital Saint-Louis ( Site 0807), Paris, Île-de-France Region
- Germany (5):
  - Klinikum Stuttgart - Katharinenhospital ( Site 0909), Stuttgart, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern ( Site 0910), Munich, Bavaria
  - Marienhospital Herne ( Site 0907), Herne, North Rhine-Westphalia
  - Universitaetsklinikum Halle ( Site 0902), Halle, Saxony-Anhalt
  - Universitaetsklinikum Jena ( Site 0903), Jena, Thuringia
- Greece (4):
  - Henry Dunant Hospital ( Site 1005), Athens, Attica
  - Metropolitan General Hospital ( Site 1001), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL ( Site 1000), Chaidari/Athens, Attica
  - European Interbalkan Medical Center-Oncology Department ( Site 1008), Thessaloniki
- Hungary (5):
  - Szegedi Tudomanyegyetem ( Site 1113), Szeged, Csongrád megye
  - Gyor- Moson- Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz ( Site 1116), Győr, Győr-Moson-Sopron
  - Heves Vármegyei Markhot Ferenc Oktatókórház és Rendelőintézet ( Site 1118), Eger, Heves County
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz Nyiregyhazi Josa Andras Tagkorhaza ( Site 1117), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Debreceni Egyetem Klinikai Kozpont ( Site 1112), Debrecen
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 1202), Milan, Lombardy
  - Istituto Nazionale Tumori Regina Elena ( Site 1201), Rome, Roma
  - Azienda USL 8 di Arezzo ( Site 1203), Arezzo
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 1200), Roma
- Netherlands (2):
  - Rijnstate ( Site 1307), Arnhem, Gelderland
  - Erasmus MC ( Site 1300), Rotterdam, South Holland
- Peru (3):
  - Oncosalud ( Site 0701), Lima, Lima Province
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 0702), San Isidro, Lima region
  - Hospital Militar Central Luis Arias Schereiber ( Site 0700), Lima
- Poland (3):
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością MEDIC-R Sp.k ( Site 1402), Poznan, Greater Poland Voivodeship
  - Szpital Wojewódzki im. Świętego Lukasza SP ZOZ w Tarnowie ( Site 1404), Tarnów, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Układu Moczowego ( Site 1401), Warszawa, Lesser Poland Voivodeship
- Spain (6):
  - Hospital Universitari Parc Tauli ( Site 1505), Sabadell, Barcelona
  - Hospital Insular de Gran Canaria ( Site 1502), Las Palmas de Gran Canaria, Canary Islands
  - Hospital Clinico San Carlos... ( Site 1500), Madrid
  - Hospital Universitario 12 de Octubre ( Site 1507), Madrid
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID ( Site 1506), Madrid
  - Hospital Universitario Virgen Macarena ( Site 1504), Seville
- Faculty of Medicine - Khon Kaen University ( Site 3001), Muang, Changwat Khon Kaen, Thailand
- United Kingdom (2):
  - St Bartholomew s Hospital ( Site 1700), London, London, City of
  - Torbay Hospital ( Site 1701), Torquay

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/